CLINICAL TRIAL: NCT05280340
Title: Advancing IL-1Ra to Prevent Inflammatory Disease in Preterm Infants - Pilot
Brief Title: Anakinra for Preterm Infants Pilot
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Monash Medical Centre (Other)
Collaborators: Monash University (Other); Hudson Institute of Medical Research (Unknown); Te Whatu Ora - Health New Zealand (Unknown); University of Auckland, New Zealand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RES 21-0000-681A
Record Dates: First submitted 2022-02-01; First posted 2022-03-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prematurity; Extreme; Inflammation
Keywords: anakinra; IL-1Ra; bronchopulmonary dysplasia; diffuse white matter injury
MeSH Terms: conditions — Premature Birth; Inflammation; Bronchopulmonary Dysplasia | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anakinra (Experimental): First 6 enrolled infants given 1.0mg/kg anakinra alternate daily IV for first 3 weeks of life.
  Remaining 18 enrolled infants given 0.8mg/kg anakinra daily IV for the first 3 weeks of life, if infant is ≥ 26 weeks gestation.
  If infant is < 26 weeks gestation, dosing of 1.0mg/kg anakinra alternate daily IV for the first 3 weeks of life, will continue (3 infants only).
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra will be given to enrolled infants starting in the first 24hrs of life for the first 3 weeks of life.
  Other Names: Kineret

SUMMARY:
Phase I/II study of anakinra to prevent the impact of perinatal inflammation in extremely premature infants.

DETAILED DESCRIPTION:
With improvements in antenatal and neonatal care over the last 20 years, now infants are born as early as 22 weeks gestation and survive to discharge from hospital. This increased survival comes with increased risk of long term issues such as cerebral palsy and chronic lung disease. There is strong evidence to show these risks are increased due to an underlying inflammatory process initiated around the time of premature birth. This study aims to prove the safety of treating infants born between 24-27+6 weeks gestation with Anakinra, a medication which is similar to an anti-inflammatory molecule the body makes itself called Interleukin 1 Receptor Antagonist (IL-1Ra). Anakinra acts to reduce the inflammatory response and is currently used in adults and children as young as 8 months to manage autoimmune inflammatory conditions. This study looks at the safety of giving Anakinra to babies born extremely premature, over the first 3 weeks of life. Once safety is established, the investigators will conduct a larger trial studying the efficacy of this treatment for reducing the risk of long-term complications caused by neonatal inflammation in extremely preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Born at 24 to 27+6 weeks gestation

Exclusion Criteria:

* Inability of the legal representatives to consent
* Any disease or condition that the investigators judge could confound the trial results; these include, but are not limited to, genetic syndromes, severe cardiac abnormalities, substantial pre-/perinatal compromise (profound/severe hypoxia (SaO2 <80% for >3h), congenital diaphragmatic hernia, intrauterine stroke and others.
* Imminent death

Ages: 24 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related serious adverse reactions (suspected and unexpected) | 3 weeks
  Monitoring of vital signs and documentation of any significant adverse effects, for the duration of treatment which is 3 weeks, such as cardiorespiratory deterioration requiring escalation of therapy (need to start or increase inotropic medication), need for cardiopulmonary resuscitation, incidence of sepsis and death within 15mins of infusion. Continuously collected physiological data will be summarised as area under the curve in 24h epochs. Serum creatinine will be monitored for incidence of acute kidney injury on days 3, 7 and 14. Liver function will be monitored for incidence of drug-induced liver injury on days 3, 7 and 14.

SECONDARY OUTCOMES:
Plasma interleukin-1 receptor antagonist levels will be measured and reported in pg/mL for each participant conferred by treatment with anakinra | 22 days
  Blood will be taken prior to commencement of the trial medication, then at 6 & 12hr post-dose on days 1 and 22 and 12hr post dose on day 3, 7 and 14 and the IL-1Ra level recorded in pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Nold, Prof, Principal Investigator — Monash University; Claudia Nold, Prof, Principal Investigator — Hudson Institute of Medical Research; Rod Hunt, Prof, Principal Investigator — Monash University; Rob Galinsky, Dr, Principal Investigator — Hudson Institute of Medical Research; Gergely Toldi, Dr, Principal Investigator — Starship Children's Hospital, Te Whatu Ora - Health New Zealand
Locations (2):
- Monash Health, Clayton, Victoria, Australia
- Starship Children's Hospital, Te Whatu Ora - Health New Zealand, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Green EA, Metz D, Galinsky R, Atkinson R, Skuza EM, Clark M, Gunn AJ, Kirkpatrick CM, Hunt RW, Berger PJ, Nold-Petry CA, Nold MF. Anakinra Pilot - a clinical trial to demonstrate safety, feasibility and pharmacokinetics of interleukin 1 receptor antagonist in preterm infants. Front Immunol. 2022 Oct 27;13:1022104. doi: 10.3389/fimmu.2022.1022104. eCollection 2022. PMID 36389766